CLINICAL TRIAL: NCT01110343
Title: Conventional Versus Mindfulness Intervention in Parents of Children With Disabilities
Brief Title: Conventional vs Mindfulness Intervention in Parents of Children With Disabilities
Acronym: PSIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Elisabeth Dykens, Director of Vanderbilt Kennedy Center, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090965; 1RC1AT005612-01 (NIH)
Record Dates: First submitted 2010-04-13; First posted 2010-04-26 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2010-04

CONDITIONS: Psychological Stress; Depression; Anxiety
Keywords: parent stress; parent coping; parent anxiety; parent health; parent depression
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mindfulness intervention group (Active Comparator): Mindfulness intervention is a formatted curriculum based on Mindfulness based stress reduction techniques which have proven effective in reducing stress related to pain, everyday living and medical and psychiatric disorders.
  Interventions: Behavioral: mindfulness intervention
- conventional parent support group (Active Comparator): a 6 week behavioral program, with weekly 1.5 hour sessions with a trained parent mentor, 3 monthly booster sessions and follow-up.
  Interventions: Behavioral: Conventional parent Support Group

INTERVENTIONS:
Behavioral: mindfulness intervention — a 6 -week behavioral intervention lasting 1.5 hours per week with a trained parent mentor, 3 monthly booster sessions and follow-up
  Arms: mindfulness intervention group
Behavioral: Conventional parent Support Group — a 6 week behavioral program, consisting of 1.5 hour weekly sessions run by a trained parent mentor with a structured curriculum based on the strengths of support groups like emotional support, advocacy and training. There are 3 monthly booster sessions and follow-up.
  Arms: conventional parent support group

SUMMARY:
This application compares the effectiveness of a conventional Parent Group intervention to Mindfulness- Based Stress Reduction (MBSR) in parents of children with autism spectrum disorders (ASD) and other disabilities. Parent groups are widely-used to provide information, emotional support, education and advocacy. MBSR is efficacious for people with medical, psychiatric or other concerns, and teaches stress reduction through mindfulness training and practice. In contrast to conventional parent groups, the investigators' studies suggest that mindfulness-based interventions may be particularly effective in reducing stress and improving the health and mental health of parents of children with disabilities. The investigators will assess parent factors that may correlate with intervention efficacy in the 2 treatment arms.

DETAILED DESCRIPTION:
Specific Aim 1. To compare the effectiveness of Parent Groups versus MBSR interventions in parents of children with ASD or other developmental disabilities.

Hypothesis 1: Mothers and fathers in both treatment groups will show reduced stress, depression, and anxiety, and increased life satisfaction, health, and well-being. Treatment effects will be more pronounced in MBSR, including more normalized diurnal cortisol patterns.

Hypothesis 2: Improved parental outcomes will persist after treatment, and relate to booster session attendance, and/or the frequency that parents practice techniques learned in each treatment. Improvements will be sustained longer in the MBSR treatment. Parental benefits will impact families, and may be associated with improved child behaviors or less family conflict.

Hypothesis 3. The composition of intervention groups in Year 2 will be adjusted based on Year 1 data, and may reflect continued separation or integration of ASD vs other disability groups, or new combinations of participants.

Specific Aim 2: To identify aspects of maternal, family or child functioning that help explain variability in responses to Parent Group or MBSR interventions.

Hypothesis 4: Mothers or fathers with relatively more stress, health or mental health problems, will show more robust treatment responses. Variability in treatment responses may be associated with child age, maternal age, family ethnicity, and child behavior problems.

Hypothesis 5. Outcomes may relate to factors in the interventionists, greater treatment responses will be found when parents are matched with peer-mentors of the same gender, ethnicity, and child diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* parent of a child with a known developmental disorder
* parent of a child with a chronic medical condition with known lifelong physical and mental effects, e.g., childhood cancer, cystic fibrosis, and muscular dystrophy

Exclusion Criteria:

* those who are not parent of a child with a known developmental disorder or medical condition

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Parenting Stress Index Scores | day 1 of week 6, active intervention phase
  Parenting Stress Index standard scores will show treatment effects of intervention by day one of week six of active intervention phase.

SECONDARY OUTCOMES:
Beck Depression Inventory, Parenting Stress Index, Epworth Sleep Scale, Positive Affect Index, Life Satisfaction Scale, Mindfulness Questionnaire, Ryff's Well being Scale, Health Questionnaire, Achenbach Child Behavior Checklist | at day 1 of week six -active intervention phase
  This standardized self report measure will determine if the treatment arms differ in effectiveness and whether overall depression symptoms are alleviated with treatment.
Beck Anxiety Inventory | at day one of week 6, active intervention phase
  This standardized measure of physiological anxiety symptoms will show treatment effects by week 6 in response to 2 different treatment arms.
Salivary Cortisol measures | at day 1 of week 6, active intervention phase
  Diurnal salivary cortisol measures will show differences to 2 arms of treatment intervention after 6 weeks of active intervention.
Ryff's scale of Well-being | on day 1 of week 6, active intervention phase
  This self report measure of well-being will show treatment effects of interventions on week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth M Dykens, PHD, Principal Investigator — Vanderbilt Kennedy Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States